CLINICAL TRIAL: NCT04482335
Title: PRECISion medicinE Across the Disease Continuum to Prevent and Treat Rheumatoid Arthritis
Acronym: PRECISE-RA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof. Maya H. Buch, Clinical Professor of Rheumatology, University of Manchester
Other Study IDs: 281253
Record Dates: First submitted 2020-04-08; First posted 2020-07-22 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A maximum of 75mls of blood may be taken to enable the range of experimental studies.
  The blood may be drawn into a combination of EDTA, lithium heparin, red clotted, citrate and PAXGENE/TEMPUS tubes, according to planned experiments at each time point. Samples will be collected fasting at specific timepoints if indicated.
  Similarly, synovial fluid may also be aspirated from a clinically inflamed joint (usually as part of clinical indication), and used for research purpose. Urine samples may also be collected (usually as part of clinical indication), and used for research purpose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Main Study: Participants complete questionnaires and agree to have their retrospective and prospective medical data used as part f this research project. All participants will take part in this arm.
  Interventions: Other: No intervention
- Biosample Sub-Study: A subset of the participants will take part of this. Participants will agree to have blood samples taken at regular intervals or at the point of a flare or when their treatment changes. They might also be asked to provide urine samples.
  Interventions: Other: No intervention
- Synovial Biopsy and Synovial Fluid Sub-Study: A subset of the participants will take part of this. Participants will agree to synovial biopsies at regular intervals or at the point of a flare or when their treatment changes. They might also be asked to donate waste synovial fluid.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The study will recruit patients referred to the Rheumatology Out-patient departments. Patients will be recruited to the study or control groups (healthy or disease controls who will be age and sex-matched) as needed. The study will first open to recruitment at Manchester University Hospitals NHS Foundation Trust and then open at other NHS Trusts. Patients will be asked to participate in longitudinal (clinical/imaging/biosample) data and/or sample collection that will improve our understanding of underlying disease mechanisms and identify improved diagnostic, prognostic and predictive biomarkers to understand progression of disease and drug response or resistance.

DETAILED DESCRIPTION:
Main Study

Consent to this ethics' main programme will permit collection of routinely collected data and use for research activities. Patients may be recruited at any point along their disease continuum (e.g. time of initial diagnosis, before/after a new treatment intervention, at time of disease flare or stable state).

Patients with established disease who are recruited to the study during their follow up appointments will have pre-existing results and clinical documentation. These retrospective data may also be collected where possible using information documented in case-notes and/or hospital information systems.

Some study-specific information will also be collected.

In addition to the main study, participants will be offered the opportunity to consent to participate in one or more sub-studies which include the additional research procedures (entitled 'basic biological' and 'synovial biopsy'). It will be possible for patients to participate in more than one sub-study.

The sub-studies aim to explore the mechanisms that may underlie change over the disease continuum, not just at disease initiation. In particular, the researchers would wish to obtain samples and imaging that coincide with a change in disease profile as well as with loss of disease control. Acquiring pre- and post-treatment blood/tissue samples and images would allow the investigation of changes in disease pathogenesis, the role of specific therapies, and identification of treatment response indicators. The researchers would therefore ask the permission of some individuals to obtain samples or images at additional time-points to coincide with events along their disease continuum.

Basic Biological sub-study

This sub-study will facilitate identification of prognostic markers of disease, mechanism and predictive markers of drug response. As part of an in-house investigation of biomarkers and mechanisms, DNA, serum, plasma, synovial joint fluid, and urine may be collected and stored. Patients will have the opportunity to consent separately to the genetic (DNA) component.

A maximum of 75mls of blood may be taken to enable the range of experimental studies. The samples will be taken at relevant clinical time points related to diagnosis, disease profile, disease activity state and/or treatment related time points; thus samples may be taken at one time point or repeated depending on the individual study objective and status of the patient.

Synovial biopsy sub-study

Patients will be asked to consent to a synovial biopsy of an affected joint to provide synovial tissue for research purposes. Synovial joint fluid may also be collected as part of the biopsy procedure. This will be performed by a trained clinician within our department by ultrasound-guidance. Depending on the research question being addressed, biopsy may be taken at time of diagnosis; or before and after starting a new drug treatment; or at time of a change in disease activity/flare (that may/may not lead to change in therapy). If repeat biopsy is taken, this is typically 3 or 6 months after starting a new therapy; or may be a later time point if evaluating for change in disease characteristics and tissue biology over time.

ELIGIBILITY:
Inclusion Criteria

1. Subject ≥ 18 years of age
2. Is capable of understanding and signing an informed consent form
3. Falls into one of the following:

   1. Pre-RA - Any musculoskeletal symptom (inflammatory and/or non-inflammatory) AND either RF and/orACPA positive.
   2. UA - Inflammatory joint symptoms (including joint pain, significant early morning stiffness and joint swelling) not fulfilling any classification criteria
   3. ERA - recent clinical diagnosis of RA EstRA - known diagnosis of RA supported by evidence of established inflammatory arthritis including but not limited to synovitis, erosion, tenosynovitis.

Exclusion Criteria

1. Age less than 18 years
2. Lack of capacity to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People with early rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
• Main study - Change in Disease Activity Score in 28 Joints (DAS28) | through to study completion, an average of 2 years
  • The Disease Activity Score (DAS) assessment is a derived measurement with differential weight given to each component. The DAS28 is calculated at every visit. The components of the DAS28 ESR score assessment are: Tender/ Painful Joint Count (28), Swollen Joint Count (28); ESR, Subject General Health VAS assessment (0-100). The components of the DAS28 CRP score assessment are: Tender/Painful Joint Count (28); Swollen Joint Count (28), CRP, and the Subject General Health VAS assessment (0-100). The DAS score ranges from 0-10 and higher scores indicate high disease activity. A DAS28 value of >5.1 indicates high disease activity, 3.2 <DAS28 ≤5.1 and DAS28 ≤3.2 are defined as moderate and low disease activity. Patients may be considered to be in remission phase if DAS28 is <2.6
• Biosample substudy - Change in serum biomarkers, gene expression and the distribution of cell populations in biological samples (peripheral blood, synovial fluid, urine) using ELISA, sequencing, flow cytometry and CyTOF | through to study completion, an average of 2 years
  • Biosample substudy - Change in serum biomarkers, gene expression and the distribution of cell populations in biological samples (peripheral blood, synovial fluid, urine) using ELISA, sequencing, flow cytometry and CyTOF
• Synovial biopsy substudy - Changes in immunological markers of inflammation in synovial tissue | Baseline +/- week 12 or 24 after change in therapy
  • Synovial biopsy substudy - Changes in immunological markers of inflammation in synovial tissue

SECONDARY OUTCOMES:
• Change in Patient reported outcome measure - Rheumatoid Arthritis Quality of Life (RAQoL) | through to study completion, an average of 2 years
  • The RAQoL questionnaire consists of 30 items. The overall score is the sum of individual item scores, with a lower score indicating better QoL (range 0-30)
• Change in Patient reported outcome measure - Health Assessment Questionnaire (HAQ) | through to study completion, an average of 2 years
  • The HAQ questions are assessed on a 4-point Likert scale (0 = without difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Total HAQ score ranges from 0-3.0 in increments of 0.125. Higher scores indicate worse functioning.
• Change in Patient reported outcome measure - EuroQoL (EQ-5D) | through to study completion, an average of 2 years
  • The EQ-5D consists of 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) rated on a 3 level scale (no problems, some or moderate problems, extreme problems). Rated levels are coded as number 1, 2 or 3 and reported as a five-digit number ranging from 11111 (no problems in all domains) to 55555 (extreme problems in all domains)
• Change in Patient reported outcome measure - Functional Assessment of Chronic Illness Therapy - fatigue (FACIT-fatigue) | through to study completion, an average of 2 years
  • FACIT-fatigue is a 13-item instrument measure of fatigue scored on a 0-4 response scale. All items are summed to create a final score (range 0-52). Higher scores indicate greater fatigue.
• Change in Patient reported outcome measure - Hospital Anxiety and Depression Scale (HADs) | through to study completion, an average of 2 years
  • HADs consists of two subscales (anxiety and depression) with a total of 14 items - each scored on a scale from 0 to 3. Total scores range from 0-21 for each subscale (0-7 = normal, 9-10 = borderline abnormal, 11-21 = abnormal)
• Change in Patient-completed visual analogue scales - pain (VAS-pain) | through to study completion, an average of 2 years
  • VAS-pain measures pain on the day on a visual analogue scale (range 0-100) with higher scores indicating worse pain
• Change in Patient-completed visual analogue scales - disease activity (VAS-DA) | through to study completion, an average of 2 years
  • VAS-DA measures the state of arthritis (swelling and stiffness) on the day on a visual analogue scale (range 0-100) with higher scores indicating extremely active arthritis
• Change in Patient-completed visual analogue scales - fatigue (VAS-fatigue) | through to study completion, an average of 2 years
  •VAS-fatigue measures overall fatigue on the day on a visual analogue scale (range 0-100) with higher scores indicating worse fatigue
• Change in Patient-completed visual analogue scales - general health (VAS-GH) | through to study completion, an average of 2 years
  • VAS-GH measures general state of health on the day on a visual analogue scale (range 0-100) with higher scores indicating poor state of health
• Change in Physician-completed visual analogue scale of disease activity | through to study completion, an average of 2 years
  • Physician-completed visual analogue scale of disease activity measures disease activity as rated by the physician on a visual analogue scale (range 0-100) with higher scores indicating extremely active disease
• Change in joint damage as measured by conventional radiography of hands and feet | through to study completion, an average of 2 years
  • Change in joint damage as measured by conventional radiography of hands and feet
• Change from baseline in Ultrasound (US) synovitis as measured by Power Doppler Ultrasound (PDUS) | through to study completion, an average of 2 years
  • Change from baseline in Ultrasound synovitis as measured by Power Doppler Ultrasound (PDUS)

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Royal Infirmary, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No